CLINICAL TRIAL: NCT03708627
Title: The Role of Bimatoprost in Graves' Periorbitopathy
Brief Title: Bimatoprost as a Treatment for Graves' Orbitopathy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00294393
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will evaluate clinical photos. Other measures such as Hertel's exophthalmometry values are objective outcomes which will be made available to the Principal Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimatoprost in more proptotic eye (Experimental): Patients instill Bimatoprost in their more proptotic eye one nightly
  Interventions: Drug: Bimatoprost Ophthalmic
- Control (No Intervention): Bimatoprost is not instilled in the patient's fellow eye

INTERVENTIONS:
Drug: Bimatoprost Ophthalmic — Bimatoprost, aka Lumigan, one drop in one eye nightly
  Arms: Bimatoprost in more proptotic eye

SUMMARY:
Testing whether Bimatoprost, a topical eye drop used for glaucoma, can be used to induce periorbital fat atrophy in patients with Graves' disease

ELIGIBILITY:
Inclusion Criteria: Graves' Ophthalmopathy with Exophthalmos/Proptosis -

Exclusion Criteria: Active Graves Disease, Currently pregnant, Taking Steroids

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in periorbital fat causing improvement in proptosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emily Li, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- University of Washington, Seattle, Washington, United States